CLINICAL TRIAL: NCT07311447
Title: The Effect of Target-Controlled Infusion (TCI) on Neurocognitive Functions in Postoperative Sedoanalgesia Management in Geriatric Patients Undergoing Major Surgery
Brief Title: Target-Controlled Infusion and Postoperative Neurocognitive Outcomes in Geriatric Patients
Acronym: TCI-NEURO
Status: Completed | Type: Observational
Sponsor: Namigar Turgut (Other)
Responsible Party: Sponsor-Investigator, Namigar Turgut, Professor of Anesthesiology and Intensive Care, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: Tascıoglu-TCI-POCD-2025
Record Dates: First submitted 2025-12-08; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Cognitive Dysfunction (POCD); Neurocognitive Function; Sedation and Analgesia; Geriatric Patients
Keywords: Target-Controlled Infusion (TCI); Manual Infusion; Geriatric Patients; Mini-Mental State Examination (MMSE)
MeSH Terms: conditions — Postoperative Cognitive Complications; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCI Group: Patients receiving postoperative sedoanalgesia with Target-Controlled Infusion (TCI). Sedation and analgesia were maintained using a target-controlled infusion system adjusted according to BIS and RASS monitoring.
- Manual Infusion Group: Patients receiving postoperative sedoanalgesia with manually adjusted infusion without TCI. Sedation and analgesia were titrated manually based on BIS and RASS monitoring.

SUMMARY:
This prospective observational study aims to evaluate the effects of target-controlled infusion (TCI) on postoperative neurocognitive function in geriatric patients undergoing major non-cardiac surgery. Elderly patients are at increased risk of postoperative cognitive dysfunction due to physiological changes and anesthesia-related factors. In this study, sedation management with TCI will be compared to manual infusion. Neurocognitive function will be assessed at multiple time points using the Mini-Mental State Examination (MMSE), and sedation levels will be monitored with the Bispectral Index (BIS) and the Richmond Agitation-Sedation Scale (RASS). The study aims to provide insights into safer sedation practices and improved cognitive outcomes in elderly surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Undergoing noncardiac, nonneurosurgical major surgery under general anesthesia
* Monitored postoperatively in the intensive care unit
* Provided informed consent to participate in the study

Exclusion Criteria:

* Cardiac or neurosurgical procedures
* Patients younger than 65 years
* Glasgow Coma Scale < 8
* No informed consent
* Body mass index (BMI) > 35
* Communication difficulties preventing cognitive testing
* Known allergy to study medications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric patients aged 65 years and older who undergo noncardiac, nonneurosurgical major surgery under general anesthesia and are monitored postoperatively in the intensive care unit. The study includes patients managed with either Target Controlled Infusion (TCI) or manual infusion for postoperative sedation and analgesia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in neurocognitive function score (Mini-Mental State Examination,MMSE) | Preoperative baseline (within 24 hours before anesthesia) to 72 hours postoperatively
  Between-group difference in the change of Mini-Mental State Examination (MMSE) total score from baseline to 72 hours after surgery, comparing target-controlled infusion (TCI) versus manual infusion. The MMSE is a widely used cognitive screening tool with a total score range of 0 to 30, where higher scores indicate better cognitive function.

SECONDARY OUTCOMES:
Total sedative and analgesic drug consumption | From admission to the intensive care unit (ICU) until completion of the postoperative sedation period (approximately 0-72 hours postoperatively).
  Total amount of sedative and analgesic medications administered during the postoperative sedation period in both groups (TCI vs manual infusion). Lower consumption may indicate more efficient sedation management.
Hospital length of stay | From the day of surgery until hospital discharge (up to 40 days).
  Total duration of hospitalization from the day of surgery until the patient is medically ready for discharge. Comparisons will be made between the TCI and manual infusion groups to evaluate whether postoperative sedation method influences overall hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Namigar Turgut, MD, Principal Investigator — İstanbul Prof. Dr. Cemil Taşcıoğlu City Hospital; Zekeriya Ervatan, MD, Study Chair — İstanbul Prof. Dr. Cemil Taşcıoğlu City Hospital
Locations (1):
- İstanbul Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and ethical restrictions.